CLINICAL TRIAL: NCT01237821
Title: A MULTI-CENTER, DOUBLE-BLIND CLINICAL TRIAL TO EVALUATE THE SAFETY AND EFFICACY OF TWO ACNE CREAMS IN SUBJECTS WITH MILD TO MODERATE ACNE VULGARIS
Brief Title: Comparing OTC Acne Treatment to Prescription Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Loreal USA (Industry)
Responsible Party: Principal Investigator, Amy Longenecker, RN, CCRC, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS1007033A
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BenzaClin (Active Comparator): Evaluate and compare tolerance and efficacy of two anti-acne creams, Effaclar and Benzaclin over a twelve week period.Inclusion- males and females ages 18-50, mild to moderate acne vulgaris with > or equal to 15 inflammatory lesions, > or equal to 20 non-inflammatory lesions, avoid excessive sun exposure or tanning beds throughout the study, . Exclusion- Participants who have another skin condition that will interfere with lesion counting or assessments
  Interventions: Drug: BenzaClin
- effaclar (Active Comparator): Evaluate and compare tolerance and efficacy of two anti-acne creams, Effaclar and Benzaclin over a twelve week period.Inclusion- males and females ages 18-50, mild to moderate acne vulgaris with > or equal to 15 inflammatory lesions, > or equal to 20 non-inflammatory lesions, avoid excessive sun exposure or tanning beds throughout the study, . Exclusion- Participants who have another skin condition that will interfere with lesion counting or assessments
  Interventions: Drug: Effaclar

INTERVENTIONS:
Drug: BenzaClin — Topical, 1% Clindamycin/5% Benzoyl Peroxide, BID, 12 weeks
  Arms: BenzaClin
Drug: Effaclar — Topical, Bid, 12 weeks
  Arms: effaclar

SUMMARY:
This research is being done to find out the safety and efficacy of two acne creams, Effaclar and Benzaclin when used twice daily with a topical retinoid. Effaclar and Benzaclin are FDA approved for the treatment of acne.

DETAILED DESCRIPTION:
There are many products on the market to treat facial acne. The medication that this study will be evaluating, Benzaclin and Retin-A have been approved by the FDA and is available by prescription, Effaclar is an over the counter product. This study will hopefully recognize a treatment combination that is effective in reducing acne vulgaris in adults 18-50.

ELIGIBILITY:
Inclusion Criteria:males and females ages 18-50, mild to moderate acne vulgaris with > or equal to 15 inflammatory lesions, > or equal to 20 non-inflammatory lesions, avoid excessive sun exposure or tanning beds throughout the study

Exclusion Criteria:Participants who have another skin condition that will interfere with lesion counting or assessments

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Oresajo, PhD, Study Director — Loreal USA
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BenzaClin: Evaluate and compare tolerance and efficacy of two anti-acne creams, Effaclar and Benzaclin over a twelve week period.
  BenzaClin: Topical, 1% Clindamycin/5% Benzoyl Peroxide, BID, 12 weeks
- Effaclar: Evaluate and compare tolerance and efficacy of two anti-acne creams, Effaclar and Benzaclin over a twelve week period.
  Effaclar: Topical, (Benzoyl peroxide 5.5%) Bid, 12 weeks
Period: Overall Study
Arm/Group | BenzaClin | Effaclar
Started | 32 | 34
Completed | 26 | 34
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BenzaClin | Effaclar | Total
Number analyzed (Participants) | 26 | 34 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 34 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.53 (9.81) | 32.41 (9.30) | 30.92 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 26 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Treatment Tolerability Assessment: Erythema
Description: Participants were assessed for Erythema on a 4-point ordinal scale where 0= none; 1= mild; 2= moderate; and 3= severe. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: Male and female 18-50 years old, mild to moderate acne vulgaris with >15 inflammatory lesions (papules/pustules) and >20 non-inflammatory lesions (black heads/white heads) on the face.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Effaclar: Effaclar: Topical, (Benzoyl peroxide 5.5%) Bid, 12 weeks
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 0.3 [0 to 3] | 0.4 [0 to 3]
  Week 2 | 0.6 [0 to 3] | 0.4 [0 to 3]
  Week 4 | 0.3 [0 to 3] | 0.4 [0 to 3]
  Week 8 | 0.1 [0 to 3] | 0.2 [0 to 3]
  Week 12 | 0.2 [0 to 3] | 0.2 [0 to 3]
  Week 16 | 0.1 [0 to 3] | 0.1 [0 to 3]

2. Primary Outcome: Treatment Tolerability Assessment: Edema
Description: Participants were assessed for Edema on a 4-point ordinal scale where 0= none; 1= mild; 2= moderate; and 3= severe. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 0.1 [0 to 3] | 0.1 [0 to 3]
  Week 2 | 0.2 [0 to 3] | 0.2 [0 to 3]
  Week 4 | 0.1 [0 to 3] | 0.2 [0 to 3]
  Week 8 | 0.0 [0 to 3] | 0.1 [0 to 3]
  Week 12 | 0.0 [0 to 3] | 0.0 [0 to 3]
  Week 16 | 0.0 [0 to 3] | 0.0 [0 to 3]

3. Primary Outcome: Treatment Tolerability Assessment: Dryness
Description: Participants were assessed for Dryness on a 4-point ordinal scale where 0= none; 1= mild; 2= moderate; and 3= severe. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 0.4 [0 to 3] | 0.2 [0 to 3]
  Week 2 | 0.9 [0 to 3] | 0.7 [0 to 3]
  Week 4 | 0.6 [0 to 3] | 0.3 [0 to 3]
  Week 8 | 0.2 [0 to 3] | 0.2 [0 to 3]
  Week 12 | 0.2 [0 to 3] | 0.2 [0 to 3]
  Week 16 | 0.0 [0 to 3] | 0.0 [0 to 3]

4. Primary Outcome: Treatment Tolerability Assessment: Peeling
Description: Participants were assessed for Peeling on a 4-point ordinal scale where 0= none; 1= mild; 2= moderate; and 3= severe. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 0.1 [0 to 3] | 0.0 [0 to 3]
  Week 2 | 0.5 [0 to 3] | 0.6 [0 to 3]
  Week 4 | 0.5 [0 to 3] | 0.3 [0 to 3]
  Week 8 | 0.1 [0 to 3] | 0.2 [0 to 3]
  Week 12 | 0.1 [0 to 3] | 0.1 [0 to 3]
  Week 16 | 0.0 [0 to 3] | 0.0 [0 to 3]

5. Primary Outcome: Facial Skin Assessment: Skin Tone (Clarity)
Description: The facial skin was assessed for skin tone (clarity) on a 10-point visual analog scale with 0 indicating a favorable rating and 9 indicating an unfavorable rating. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 5.3 [0 to 9] | 5.0 [0 to 9]
  Week 2 | 4.6 [0 to 9] | 4.4 [0 to 9]
  Week 4 | 4.1 [0 to 9] | 3.9 [0 to 9]
  Week 8 | 3.3 [0 to 9] | 3.2 [0 to 9]
  Week 12 | 2.6 [0 to 9] | 2.3 [0 to 9]
  Week 16 | 2.7 [0 to 9] | 2.7 [0 to 9]

6. Primary Outcome: Facial Skin Assessment: Skin Smoothness
Description: The facial skin was assessed for skin smoothness on a 10-point visual analog scale with 0 indicating a favorable rating and 9 indicating an unfavorable rating. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 5.0 [0 to 9] | 4.9 [0 to 9]
  Week 2 | 4.7 [0 to 9] | 4.5 [0 to 9]
  Week 4 | 4.2 [0 to 9] | 3.5 [0 to 9]
  Week 8 | 3.2 [0 to 9] | 2.7 [0 to 9]
  Week 12 | 2.3 [0 to 9] | 2.1 [0 to 9]
  Week 16 | 2.2 [0 to 9] | 2.3 [0 to 9]

7. Primary Outcome: Facial Skin Assessment: Skin Brightness
Description: The facial skin was assessed for skin brightness on a 10-point visual analog scale with 0 indicating a favorable rating and 9 indicating an unfavorable rating. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 5.1 [0 to 9] | 4.6 [0 to 9]
  Week 2 | 4.6 [0 to 9] | 4.1 [0 to 9]
  Week 4 | 4.0 [0 to 9] | 3.6 [0 to 9]
  Week 8 | 3.2 [0 to 9] | 2.8 [0 to 9]
  Week 12 | 2.5 [0 to 9] | 2.4 [0 to 9]
  Week 16 | 2.6 [0 to 9] | 2.6 [0 to 9]

8. Primary Outcome: Facial Skin Assessment: Appearance of Pores
Description: The facial skin was assessed for the appearance of pores on a 10-point visual analog scale,with 0 indicating a favorable rating and 9 indicating an unfavorable rating. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 4.6 [0 to 9] | 4.6 [0 to 9]
  Week 2 | 4.3 [0 to 9] | 4.5 [0 to 9]
  Week 4 | 4.1 [0 to 9] | 4.2 [0 to 9]
  Week 8 | 3.5 [0 to 9] | 3.6 [0 to 9]
  Week 12 | 3.2 [0 to 9] | 3.1 [0 to 9]
  Week 16 | 3.1 [0 to 9] | 3.3 [0 to 9]

9. Primary Outcome: Facial Skin Assessment: Overall Appearance
Description: The facial skin was assessed for overall appearance on a 10-point visual analog scale with 0 indicating a favorable rating and 9 indicating an unfavorable rating. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 5.1 [0 to 9] | 5.0 [0 to 9]
  Week 2 | 4.7 [0 to 9] | 4.4 [0 to 9]
  Week 4 | 4.3 [0 to 9] | 3.9 [0 to 9]
  Week 8 | 3.2 [0 to 9] | 3.1 [0 to 9]
  Week 12 | 2.6 [0 to 9] | 2.4 [0 to 9]
  Week 16 | 2.5 [0 to 9] | 2.6 [0 to 9]

10. Primary Outcome: Facial Skin Assessment: Global Acne Assessment
Description: The facial skin was assessed for global acne assessment on a 10-point visual analog scale with 0 indicating a favorable rating and 9 indicating an unfavorable rating. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 3.4 [0 to 9] | 3.1 [0 to 9]
  Week 2 | 3.1 [0 to 9] | 2.7 [0 to 9]
  Week 4 | 2.5 [0 to 9] | 2.3 [0 to 9]
  Week 8 | 2.2 [0 to 9] | 2.1 [0 to 9]
  Week 12 | 1.7 [0 to 9] | 1.7 [0 to 9]
  Week 16 | 2.2 [0 to 9] | 2.0 [0 to 9]

11. Primary Outcome: Facial Lesion Counts: Open Comedones
Description: Participants were assessed for facial open comedomes and the total number present was recorded. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: Open Comedone Count
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
Open Comedone Count
  Baseline | 8.4 [1 to 24] | 8.3 [1 to 24]
  Week 2 | 5.3 [1 to 12] | 4.8 [1 to 12]
  Week 4 | 3.2 [1 to 12] | 3.6 [1 to 12]
  Week 8 | 2.9 [1 to 9] | 3.5 [1 to 9]
  Week 12 | 1.3 [0 to 5] | 0.9 [0 to 5]
  Week 16 | 2.0 [0 to 5] | 0.8 [0 to 5]

12. Primary Outcome: Facial Lesion Counts: Closed Comedones
Description: Participants were assessed for facial closed comedomes and the total number present was recorded. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: Closed Comedone Count
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
Closed Comedone Count
  Baseline | 22.5 [5 to 38] | 23 [5 to 38]
  Week 2 | 16.0 [5 to 24] | 14.8 [7 to 22]
  Week 4 | 9.8 [1 to 15] | 13.7 [1 to 17]
  Week 8 | 8.3 [1 to 21] | 9.8 [1 to 14]
  Week 12 | 6.4 [0 to 11] | 8.4 [0 to 15]
  Week 16 | 9.4 [0 to 12] | 10.0 [0 to 17]

13. Primary Outcome: Facial Lesion Counts: Papules
Description: as for outcome 11
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: Papule Count
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
Papule Count
  Baseline | 17.4 [6 to 26] | 15.7 [4 to 25]
  Week 2 | 12.0 [2 to 19] | 9.0 [3 to 14]
  Week 4 | 8.0 [1 to 16] | 6.6 [1 to 10]
  Week 8 | 6.4 [1 to 9] | 5.8 [1 to 9]
  Week 12 | 5.3 [1 to 9] | 4.0 [1 to 7]
  Week 16 | 6.8 [1 to 11] | 4.5 [1 to 7]

14. Primary Outcome: Facial Lesion Counts: Pustules
Description: Participants were assessed for facial pustules and the total number present was recorded. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: Pustules Count
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
Pustules Count
  Baseline | 3.6 [0 to 8] | 3.9 [0 to 8]
  Week 2 | 2.3 [0 to 8] | 1.4 [0 to 5]
  Week 4 | 1.4 [0 to 5] | 1.3 [0 to 5]
  Week 8 | 0.8 [0 to 4] | 0.9 [0 to 4]
  Week 12 | 0.5 [0 to 4] | 0.5 [0 to 4]
  Week 16 | 1.0 [0 to 4] | 1.7 [0 to 5]

15. Primary Outcome: Facial Lesion Counts: Noninflammatory Lesions
Description: Participants were assessed for facial noninflammatory lesions and the total number present was recorded. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: Noninflammatory Lesion Count
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
Noninflammatory Lesion Count
  Baseline | 30.9 [6 to 61] | 31.3 [10 to 65]
  Week 2 | 21.3 [5 to 48] | 19.6 [5 to 48]
  Week 4 | 13.0 [2 to 26] | 17.3 [4 to 31]
  Week 8 | 11.2 [0 to 17] | 13.3 [0 to 20]
  Week 12 | 7.7 [0 to 11] | 9.3 [0 to 21]
  Week 16 | 11.4 [0 to 19] | 10.9 [0 to 22]

16. Primary Outcome: Facial Lesion Counts: Inflammatory Lesions
Description: Participants were assessed for facial inflammatory lesions and the total number present was recorded. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: Inflammatory Lesion Count
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
Inflammatory Lesion Count
  Baseline | 21.0 [6 to 32] | 19.6 [5 to 27]
  Week 2 | 14.3 [5 to 22] | 10.4 [2 to 14]
  Week 4 | 9.4 [2 to 16] | 7.9 [2 to 15]
  Week 8 | 7.2 [0 to 12] | 6.7 [0 to 10]
  Week 12 | 5.8 [0 to 8] | 4.4 [0 to 6]
  Week 16 | 7.7 [0 to 12] | 6.2 [0 to 9]

17. Primary Outcome: Facial Lesion Counts: Total Lesion
Description: Participants were assessed for all facial lesions and the total number present was recorded. Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: Total Lesion Count
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
Total Lesion Count
  Baseline | 51.9 [12 to 66] | 51.0 [18 to 72]
  Week 2 | 35.6 [10 to 59] | 30.0 [8 to 48]
  Week 4 | 22.5 [10 to 48] | 25.1 [13 to 56]
  Week 8 | 18.5 [2 to 31] | 20.0 [5 to 25]
  Week 12 | 13.5 [2 to 22] | 13.7 [3 to 27]
  Week 16 | 19.0 [5 to 34] | 17.0 [2 to 32]

18. Primary Outcome: Subjective Tolerability of Irritation Assessment (Participant Assessed): Stinging
Description: Irritation stinging was subjectively reported by participants and captured on a 4 point ordinal scale (0= none; 1= mild; 2= moderate; 3= severe). Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 0.1 [0 to 3] | 0.0 [0 to 3]
  Week 2 | 0.8 [0 to 3] | 0.8 [0 to 3]
  Week 4 | 0.4 [0 to 3] | 0.4 [0 to 3]
  Week 8 | 0.3 [0 to 3] | 0.5 [0 to 3]
  Week 12 | 0.2 [0 to 3] | 0.3 [0 to 3]
  Week 16 | 0.1 [0 to 3] | 0.2 [0 to 3]

19. Primary Outcome: Subjective Tolerability of Irritation Assessment (Participant Assessed): Tingling
Description: Irritation tingling was subjectively reported by participants and captured on a 4 point ordinal scale (0= none; 1= mild; 2= moderate; 3= severe). Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 0.1 [0 to 3] | 0.0 [0 to 3]
  Week 2 | 0.8 [0 to 3] | 0.8 [0 to 3]
  Week 4 | 0.4 [0 to 3] | 0.4 [0 to 3]
  Week 8 | 0.3 [0 to 3] | 0.5 [0 to 3]
  Week 12 | 0.2 [0 to 3] | 0.3 [0 to 3]
  Week 16 | 0.1 [0 to 3] | 0.2 [0 to 3]

20. Primary Outcome: Subjective Tolerability of Irritation Assessment (Participant Assessed): Itching
Description: Irritation itching was subjectively reported by participants and captured on a 4 point ordinal scale (0= none; 1= mild; 2= moderate; 3= severe). Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 0.2 [0 to 3] | 0.1 [0 to 3]
  Week 2 | 0.5 [0 to 3] | 0.5 [0 to 3]
  Week 4 | 0.4 [0 to 3] | 0.4 [0 to 3]
  Week 8 | 0.3 [0 to 3] | 0.3 [0 to 3]
  Week 12 | 0.2 [0 to 3] | 0.3 [0 to 3]
  Week 16 | 0.1 [0 to 3] | 0.3 [0 to 3]

21. Primary Outcome: Subjective Tolerability of Irritation Assessment (Participant Assessed): Burning
Description: Irritation burning was subjectively reported by participants and captured on a 4 point ordinal scale (0= none; 1= mild; 2= moderate; 3= severe). Assessments were made at baseline and weeks, 2, 4, 8, and 12, with the regression phase assessment at week 16.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Effaclar | Benzaclin
Number analyzed (Participants) | 26 | 34
score on a scale
  Baseline | 0.2 [0 to 3] | 0.1 [0 to 3]
  Week 2 | 1.1 [0 to 3] | 1.0 [0 to 3]
  Week 4 | 0.6 [0 to 3] | 0.4 [0 to 3]
  Week 8 | 0.5 [0 to 3] | 0.5 [0 to 3]
  Week 12 | 0.3 [0 to 3] | 0.4 [0 to 3]
  Week 16 | 0.0 [0 to 3] | 0.1 [0 to 3]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Effaclar | BenzaClin
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/34
Other Adverse Events (participants affected / at risk) | 0/26 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No